CLINICAL TRIAL: NCT02112617
Title: Phase II Study of Proton Radiation Therapy for Neuroblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin X. Liu, MD, DPHIL, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-443
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma; Ganglioneuroblastoma
Keywords: Neuroblastoma; Childhood neuroblastoma; Ganglioneuroblastoma; Pediatric neuroblastoma
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroblastoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Radiation Therapy (PBRT) (Experimental): Proton radiation will be delivered daily for 3-4 weeks, depending on the dose prescribed by study doctor. Treatment is delivered (Monday - Friday) for 5 days (no weekends or holidays). Each treatment the participant will lie on a table for 30-45 minutes.
  Interventions: Radiation: Proton Beam Radiation Therapy

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy — Proton radiation will be delivered daily for 3-4 weeks, depending on the dose prescribed by study doctor. Treatment is delivered (Monday - Friday) for 5 days (no weekends or holidays). Each treatment the participant will lie on a table for 30-45 minutes.

SUMMARY:
This research study is evaluating a therapy called proton beam radiation therapy (PBRT) as a possible treatment for neuroblastoma.

Neuroblastoma most commonly occurs in and around the adrenal glands, which are located at the top of the kidneys. However, it can also occur in other areas where groups of nerve cells exist, such as other areas of the abdomen, neck and near the spine.

Conventional radiation therapy with photons is used as standard treatment for many patients with neuroblastic tumors. In this research study, the investigators are looking at another type of radiation called proton radiation which is known to spare surrounding tissues and organs from unnecessary radiation. Proton radiation delivers radiation to the area requiring radiation. This may reduce side effects that patients would normally experience with standard radiation therapy or other means of delivering proton radiation therapy.

In this research study, the investigators are evaluating the effectiveness of using proton radiation delivered to reduce side effects associated with radiation treatment. The investigators will also be assessing the late side effects experienced by participants in each treatment group.

DETAILED DESCRIPTION:
Proton radiation will be delivered daily for 3-4 weeks, depending on the dose prescribed by study doctor. Treatment is delivered (Monday - Friday) for 5 days (no weekends or holidays). Each treatment the participant will lie on a table for 30-45 minutes.

The radiation therapy will be outpatient at Massachusetts General Hospital.

During radiation therapy, the participant will have the following weekly assessments and procedures:

* Physical Exam
* Assess for any side effects
* Routine blood tests (weekly or at least every other week)

Post-treatment Follow Up Visit (s):

The participant will be asked to return to the clinic 3-6 months after their last dose of radiation therapy and then annually for up to 5 years for the following procedures:

* Medical History
* Physical Exam
* Diagnostic Imaging
* Assess for side effects
* Lung Function Tests (if required)
* MUGA or ECHO (if required)

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed neuroblastoma or ganglioneuroblastoma or elevated urinary catecholamine metabolites. If tumor tissue was obtained, pathological review of surgical specimen at the Massachusetts General Hospital or other DF/HCC institution is required, but preliminary report only required prior to enrollment. If no tumor tissue was obtained, urinary catecholamine metabolites are required.
* Participants do not need to have measurable disease at the time of radiation. Age ≥ 3 and ≤ 25 years at the time of diagnosis because this study evaluates this disease entity in the pediatric population which may differ from the adult population.
* Life expectancy of greater than 12 months.
* ECOG performance status ≤2 (Karnofsky ≥60%, Lansky ≥60%, see Appendix A).
* Diagnostic Imaging MRI and/or CT of the area to be treated within 8 weeks of any treatment. Baseline bone marrow biopsy and bone scan (with 99mTc-diphosphonate or MIBG scan (131I-MIBG or 123I-MIBG) from time of original diagnosis is required.
* Because radiation is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability of the patient or the patient's legal guardian to understand and the willingness to sign a written informed consent document.
* Participants or their legal guardian must sign consent prior to the initiation of radiation therapy.

Exclusion Criteria:

* Patients will be ineligible if any prior therapeutic radiation therapy > 500 cGy has been delivered.
* Patients will be ineligible if chemotherapy was completed ≥ 1 year from the planned start date of radiation therapy or if the patient is referred for radiation therapy after a relapse following a regimen with chemotherapy alone.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Pregnant females are excluded. Women of childbearing age/menstruating must have a negative pregnancy test prior to initiation of radiation therapy.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2026-06-30 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Describe late complications of radiation therapy delivered with proton radiotherapy in place of photon radiation for patients with neuroblastoma | 5 years
  To describe late complications of radiation therapy delivered with proton radiotherapy in place of photon radiation for patients with neuroblastoma. Specifically, cardiac, pulmonary, gastrointestinal, endocrine, growth and second malignancies will be described.
To evaluate acute and subacute toxicities of proton radiotherapy in place of photon radiation for patients with neuroblastoma. | 5 years
  To evaluate acute and subacute toxicities of proton radiotherapy in place of photon radiation for patients with neuroblastoma. Specifically, nausea, vomiting, diarrhea, radiation pneumonitis and skin toxicity will be described.

SECONDARY OUTCOMES:
Progression free survival | 10 years
Overall survival rates | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M. MacDonald, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States